CLINICAL TRIAL: NCT02159651
Title: Specified Drug Use-results Survey for Long-term Use of Prograf Capsules in Patient With Interstitial Pneumonia Associated With Polymyositis/Dermatomyositis
Brief Title: A Survey for Long-term Use of Prograf Capsules in Patient With Interstitial Pneumonia
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: PRGI01; 506-MA-PRGI-01 (Other: Japan Medical Affairs)
Record Dates: First submitted 2014-06-06; First posted 2014-06-10 (Estimated); Last update posted 2024-10-22 (Actual); Status verified 2020-04

CONDITIONS: Interstitial Pneumonia Associated With Polymyositis/Dermatomyositis
Keywords: tacrolimus; interstitial pneumonia; prograf
MeSH Terms: conditions — Dermatomyositis; Lung Diseases, Interstitial | interventions — Tacrolimus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Dermatomyositis group: patients with interstitial pneumonia associated with dermatomyositis
  Interventions: Drug: tacrolimus
- 2: Polymyositis group: patients with interstitial pneumonia associated with polymyositis
  Interventions: Drug: tacrolimus

INTERVENTIONS:
Drug: tacrolimus — oral
  Other Names: FK506; Prograf

SUMMARY:
This study is to evaluate the safety and the efficacy of Prograf in patients with interstitial pneumonia associated with polymyositis / dermatomyositis in acute clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patient
* Patient diagnosed with Interstitial pneumonia associated with polymyositis/dermatomyositis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with interstitial pneumonia associated with polymyositis/dermatomyositis who treated with Prograf
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to three years

SECONDARY OUTCOMES:
Respiratory function test value (%FVC, %DLco) | Up to three years
  Respiratory function is evaluated by % FVC ( percent-predicted forced vital capacity) amd %DLco (diffusion capacity of CO).
Arterial blood gas analysis value (PaO2, AaDO2) | Up to three years
  Arterial blood gas analysis by PaO2 (arterial O2 pressure) and AaDO2 (alveolar-arterial oxygen difference)
Chest CT findings | Up to three years
  CT: computed tomography
Serum KL-6 value (serum SP-D value) | Up to three years
  KL-6 (sialylated carbohydrate antigen KL-6) and SP-D (surfactant protein D) are used as marker of interstitial pneumonia
Patient disposition | Up to three years
  patient disposition includes 1)number of case report forms collected, 2)number of patients analyzed for safety, 3)number of patients analysed for efficacy
Safety assessed by the incidence of adverse events | Up to three years
  Any adverse events which include adverse events leading to death, white blood cell count, erythrocyte sedimentation rate and other abnormal findings from laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kansai
  - Kanto
  - Kyushu
  - Shikoku
  - Tōhoku

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Kuwana M, Wakasugi N, Furuya T, Uno S, Suda T. Tacrolimus in Patients With Interstitial Pneumonia Associated With Polymyositis or Dermatomyositis: Interim Report of Postmarketing Surveillance in Japan. J Rheumatol. 2022 Jul;49(7):707-718. doi: 10.3899/jrheum.210322. Epub 2022 Apr 15. PMID 35428708